CLINICAL TRIAL: NCT00709501
Title: Disseminating Effective Habits for Long-Term Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Christopher N. Sciamanna, Professor of Medicine and Public Health Sciences, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 28160
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Overweight; Obesity
Keywords: weight loss; obesity; overweight
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants in the intervention condition are encouraged to access the Achieve Together website at least once each week. During each login, the following activities will occur:
  1. Users will enter their weight and height, how well their plan for a healthy weight has been going, and clarify their goal weight.
  2. Users will answer questions about each habit they are using to lose weight
  3. Users will receive automated feedback about each habit and will be encouraged to change or delete habits that are being used but not helpful, more consistently use habits that are helpful but not used being used and to continue to use habits that are helpful and being used consistently.
  4. Users are encouraged to search for habits that have helped people of similar age and gender to themselves.
  Interventions: Behavioral: Disseminating Effective Habits for Long-term Weight Loss; Behavioral: Achieve Together website
- 2 (No Intervention): Participants in the control condition will have to wait 12 weeks before accessing the Achieve Together website. These participants will be a given a log where they can document weekly weight measurements (this part did not happen).

INTERVENTIONS:
Behavioral: Disseminating Effective Habits for Long-term Weight Loss — Comparison of weight change among those participants in the weight loss intervention (immediate access to the weight loss website) and those participants in the control group (delayed access to the weight loss website).
  Arms: 1
Behavioral: Achieve Together website — access to the Achieve Together website immediately (Arm 1) or delayed (Arm 2)
  Arms: 1

SUMMARY:
The purpose of the study is to determine whether using a web-based weight loss website can help overweight individuals lose weight.

DETAILED DESCRIPTION:
Overweight and obesity are serious threats to public health. Over the last 20 years, the percentage of overweight and obese Americans, as well as the rate of diabetes, have grown tremendously (Cowie, Rust et al. 2006).

Few individuals are successful at long-term weight loss. Long-term weight loss is an elusive, yet sought after goal for many Americans (2000). Fewer than 5% of adults are successful in maintaining a 20 pound weight loss for at least 2 years (Klem, Wing et al. 1997). While medications can be effective, they produce only small amounts of weight loss, carry a significant cost and appear to be effective only while being taken (2000). Surgery is an effective option, though the procedure has tremendous costs and potential complications (2000). This points to the need for innovative and effective treatments that helps individuals over the longer-term.

Some, but not all, web-based treatments for weight loss have been shown to be effective. A recent study by Tate and colleagues showed that individuals who received counseling emails from a human or automated emails from a computer lost more weight than individuals who received neither(7.3 kg lost v. 4.9 kg and 2.6 kg, respectively) (Tate, Jackvony et al. 2006) (Tate, Jackvony et al. 2003). The feedback in the emails was based on diet and physical activity information that the individuals entered online. Dr. Harvey-Berino and colleagues has shown that social support delivered via the Internet can help weight loss efforts to the same degree as in person support (Harvey-Berino, Pintauro et al. 2004). Other studies have been mixed in their effects (Williamson, Walden et al. 2006) (Gold, Burke et al. 2007) (Wing, Tate et al. 2006), though there has generally been an effect from human feedback delivered via a computer. Other than the recent study by Tate and colleagues, no fully automated website has been effective at producing weight loss. It is our belief that fully automated systems are needed to meet the needs, in a cost-effective manner, of the 80 million overweight Americans who will need life-long help in losing weight and in maintaining their weight loss.

During an earlier phase of the study, 50 in-depth interviews were conducted with individuals who have been successful at losing weight and keeping it off. These individuals were asked specifically about which habits they use to maintain their weight loss, how these habits are implemented and how barriers to using these habits are overcome. These interviews were transcribed and the data entered into a website, to be used as part of the intervention to be tested in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* BMI 27-40 kg/m2
* Fluently speaks and reads English
* Access to the Internet at home or at work
* Valid email address
* Access to a scale for weekly weigh-ins
* Agree not to seek additional weight loss treatment
* Agree to come back regardless of amount of weight lost
* Participant in NCT00377208

Exclusion Criteria:

* Current, planned, or previous pregnancy within 12 months
* Planned or past weight loss surgery
* Recent weight loss of >= 15 lbs in the past 6 months
* History of:

  * Myocardial infarction
  * Stroke
  * Type 1 and Type 2 diabetes
  * Unstable angina
  * Congestive heart failure
  * Inability to exercise due to severe arthritis or other musculoskeletal problems
  * Cancer (except non-melanoma skin cancer)
* Evidence of severe cognitive impairment or major psychiatric illness
* Plans to move in the next 6 months
* Answering yes to any question on the Physical Activity Readiness Questionnaire (PAR-Q)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Body weight | 3 months
  Weight will be measured using a calibrated, digital scale
Blood Pressure Control | 3-Months

SECONDARY OUTCOMES:
Physical Activity, using the International Physical Activity Questionnaire | 3 months
  Results are still being analyzed
Block 2005 FFQ for assessment of diet and physical activity | 3 Months
IWQOL-Lite, a validated, 31-item, self-report measure of obesity-specific | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N Sciamanna, M.D., MPH, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine General Clinical Research Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Kraschnewski JL, Stuckey HL, Rovniak LS, Lehman EB, Reddy M, Poger JM, Kephart DK, Coups EJ, Sciamanna CN. Efficacy of a weight-loss website based on positive deviance. A randomized trial. Am J Prev Med. 2011 Dec;41(6):610-4. doi: 10.1016/j.amepre.2011.08.012. PMID 22099238